CLINICAL TRIAL: NCT01508039
Title: A Randomised, Double-blind,Single-dose,Placebo and Single-blind Active Controlled Cross-over Study in Healthy Volunteers to Access in Effects of Intranasal Chitin Micro-particles on the Release of Cytokines From Nasal Mucosa
Brief Title: Immunological Effects From Intranasal Chitin Micro-Particles
Acronym: INCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: CMP Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMP-001-008
Record Dates: First submitted 2011-10-24; First posted 2012-01-11 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Intranasal; Chitin Micro-particles; Immunological Effects; Nasal mucosa; Cytokines; Immunological Effects from Intranasal Chitin Micro-Particles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with chitin micro-particles (Experimental): The study will involve 14-healthy subjects confirming to the inclusion criteria randomised to the treatments.
  Interventions: Other: Chitin Micro Particle

INTERVENTIONS:
Other: Chitin Micro Particle — The total spray volume for each application is 0.4 ml equivalent to a total single-dose for chitin of 2 mg (0.5 mg per 0.1 ml spray).
  A total single-dose for LPS, of 2 mg of endotoxin from Enterobacter agglomerans (0.5 mg per 0.1 ml spray)
  Other Names: Chitin micro-particle

SUMMARY:
The purpose of the study is:

* To investigate whether chitin can effect healthy adults, the nasal mucosa in a direction that will enhance the immune response to infection
* To investigate whether chitin influence of the nasal mucosa is well tolerated, and that there is no inflammation, as it seen with exposure to endotoxin.

DETAILED DESCRIPTION:
STUDY SYNOPSIS Objectives

Primary

•To assess the effects of intranasal dosing of chitin micro-particles on nasal mucosa responses with respect to the concentration of cytokines (TNF-alfa, IFN-gamma, IL-1b, IL-4 IL5, IL, 6, IL-8, IL-10 and IL-13) in nasal lavage fluid compared to dosing with placebo.

Secondary

* To assess the effects of intranasal dosing of chitin micro-particles on nasal mucosa responses with respect to the concentration of cytokines (TNF-alfa, IFN-gamma, IL-1b, IL-4 IL5, IL, 6, IL-8, IL-10 and IL-13) in nasal lavage fluid compared to dosing with active control.
* To assess the total eosinophil counts and cysteinyl leukotriene concentration in nasal lavage fluid at 4 and 8 hours post-dosing compared to pre-dosing.
* To assess the total nasal symptom scores at 4 and 8 hours post-dosing.
* To assess the safety and tolerability of chitin micro-particles dosed intranasally.

Study design

This study is a single-dose, doubled-blind placebo and single-blind active controlled 3-period cross-over study with a 2-week washout in between each treatment. The subjects will be divided into 2-groups for the study and randomised to receive a single-dose of either intranasal chitin micro-particles or placebo for the first two periods and a single dose of an active control article, lipopolysaccharide (LPS), for the third period. The treatment for the first two periods will be double-blinded and the treatment for the third period with LPS will be single-blinded.

Each single dose application for chitin micro-particles (cmp), placebo and the active control article, LPS, is to comprise two 0.1 ml metered sprays into each nostril. The total spray volume for each application is 0.4 ml equivalent to a total single-dose for chitin of 2 mg (0.5 mg per 0.1 ml spray), and a total single-dose for LPS, of 2 mg of endotoxin from Enterobacter agglomerans (0.5 mg per 0.1 ml spray).

The climate chamber where the dosing is to be performed will run at 22°C with 3.5-4 air changes per hour with clean HEPA-filtered air at a relative humidity (RH) of 35-40%

Study population

The study will involve 12-healthy subjects conforming to the inclusion criteria randomised to the treatments. The duration of each subject's participation will be c.42-days with eight visits including screening and safety follow-up.

Treatment plan and methods The study is to comprise three cross-over treatment periods, where each subject (12 in total) will receive single-doses of cmp, placebo or LPS (active control) in each of the three treatment periods. The study has been designed such that LPS is to be dosed in the last period so as to mitigate any potential issues with carry-over.

Screening is to take place in a period of c.2-6-weeks prior to dosing. After obtaining informed consent, each subject will undergo a screening visit in order to review the inclusion/exclusion criteria and confirm eligibility. Each subject will then be assigned to one of two dosing groups (6 subjects per group) for each of the three study periods in order to co-ordinate dosing at the Clinic. The initial screening will identify 4-8 additional subjects (total up to 20 screened) who will be included only if one of the originally randomized subjects drop out of the study. Subjects that are replaced will be randomized for treatment and will be required to undergo all three treatment periods.

For period 1, on day 0, the first dosing group will be randomized to receive either cmp or placebo. Subjects will be admitted to the Clinic at 8:30h to acclimatize, receive pre-dosing clinical assessment and confirm eligibility. Dosing is to start at 10:00h with assessment conducted in accordance with the procedures defined below. Subjects will remain in the Clinic until c. 20:00h. On the following day (day 1), the same subjects will receive a telephone interview safety follow-up. On day 2, the second dosing group will be randomized to receive either cmp or placebo, again receiving a telephone interview safety follow-up on following day (day 3). For period 2, on day 14, the first dosing group will receive the dose not previously assigned, either cmp or placebo and will receive a telephone interview safety follow-up the following day (day 15). On day 16, the second dosing group will also receive the dose not previously assigned, either cmp or placebo and again will receive a telephone interview safety follow-up the following day (day 17). For period 3, LPS will be dosed to the first dosing group on day 28 and to the second dosing group on day 30; with a telephone interview safety follow-up on days 29 and 31 respectively.

Following the last dosing visit, subjects will receive an end-of-study safety assessment by telephone interview on day 42 (+/- 2 days), which will include adverse events checks.

Each subject will be required to provide 10 ml of blood for haematological assessment at screening and at treatment periods 1, 2 and 3. A total of 40 ml of blood will be drawn for each subject for the entire duration of the study.

Pre-dosing

1. Safety assessment in terms of physical examination, including mouth, nose and lungs
2. Symptom questionnaire
3. Blood drawn for haematological tests
4. Nasal lavage by the nasal olive test with the persons sitting with their head bent forward for 60 seconds performed

   Post-dosing
5. Measurement of nasal symptom scores at 4 and 8-hours
6. Acoustic rhinometry test performed at 4 and 8-hours
7. Nasal lavage by the nasal olive test with the persons sitting with their head bent forward for 60 seconds performed at 4 and 8-hours
8. Symptom questionnaire performed at 4 and 8-hours
9. Safety monitoring: vital signs, heart rate, blood pressure performed at 2, 6-hours
10. Follow-up safety interview performed 24-hours after dosing (following day) which includes adverse events recording and concomitant medication check.

Primary End-point Changes in levels (maximum concentration) of TNF-alfa, IFN-gamma, IL-1b, IL-4, IL5, IL-6, IL-8, IL-10 and IL-13 in nasal lavage samples following intranasal dosing with cmp compared to placebo.

Secondary End-point Changes in levels (maximum concentration) of TNF-alfa, IFN-gamma, IL-1b, IL-4, IL5, IL-6, IL-8 IL-10 and IL-13 in nasal lavage samples following intranasal dosing with cmp compared to lipopolysaccharide active control.

Change from baseline:

1. the total eosinophil counts and cysteinyl leukotriene concentration in nasal lavage fluid following intranasal dosing with cmp
2. total nasal symptom scores at 4 and 8-hours following intranasal dosing with cmp

Safety will be assessed using the adverse events, vital signs and nasal acoustic rhinometry following dosing with cmp versus placebo.

Statistical Assessment For the cytokines and cell counts the concentrations are measured, and the log-transformed data analyzed with an ANOVA model including study day and exposure as fixed factor and participants as a random factor. These variables are described by the geometric mean, coefficient of variance (CV), relative difference between exposures including 95% confidence interval (CI), and p-value.

Because of ceiling and flooring problems in the data, heterogeneity in the (within participant) variation, or violations of the assumption of normally distributed data, it is not appropriate to analyze all the data of the outcomes like the symptom scores (change from baseline) with ANOVAs. Here non-parametric tests will be applied. A Wilcoxon Rank sum test will be used to compare the groups.

Subjective symptoms at baseline are described by the median and the inter quartile range. The data for 'change in nasal scores' are described by box-plots. The upper adjacent value in the plots is the largest data-point smaller than 75th percentile plus 3/2 times the inter quartile range. The lower adjacent value is defined in the similar way.

To compare placebo and the cmp exposure and taking into account a possible 'learning effect' the data will be analysed by a standard technique taking into account the design (cross-over). The participants will be divided into two groups due to the two possible exposure orders; one group consisting of participants having been exposed to placebo exposure before the cmp exposure; and another group of participants having been exposed to cmp before the placebo exposure. The hypothesis of no difference between cmp and placebo exposure will be tested by comparing the two groups with respect to the differences between the first and the second measurement. A Wilcoxon Rank sum test is used to compare the two groups. In a similar way we will test the hypothesis of 'no effect of learning'.

ELIGIBILITY:
Inclusion Criteria:

• healthy non-smoking male or female volunteers between 18 and 30 years of age, inclusive (at screening).

Subjects:

* asymptomatic at screening as characterized by normal appearing nasal mucosa with no active allergic rhinitis.
* be free from clinically significant cardiac, pulmonary, gastrointestinal, hepatic, neurological and psychiatric disease as determined by medical history, physical examination and screening investigations.
* with no clinically-significant deviation outside the normal ranges for blood pressure and pulse measurements.
* capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* be available to complete the study.
* satisfy a medical examiner about their fitness to participate in the study.
* provide oral and written informed consent to participate in the study.

Exclusion Criteria:

Subjects with:

* atopy
* perennial rhinitis.
* upper respiratory tract infection within 2 weeks of the first dose of study medication.
* medical conditions likely to affect the outcome of the study in the opinion of the investigator.
* nasal conditions likely to affect the outcome of the study in the opinion of the investigator, i.e. nasal septal perforations, nasal polyps, sinus disease, chronic nasal obstruction, or other nasal diseases.
* presence of any respiratory disease other than a history of mild stable asthma not requiring treatment and associated with normal lung function (defined as ≥ 80% predicted for height and age, "Danish Society of Lung Physicians 1986").
* a history of immunotherapy in the past 3 years or currently on an immunotherapy treatment course including inhaled or local corticosteroids in the past 28 days.
* any infirmity, disability, or geographic location which, in the opinion of the chief investigator, would limit compliance with the protocol.
* infection of the upper airways/lower airways, sinus, or ear, including viral infections in the 14 days prior to screening and at the start of/or during the treatment period.
* subjects with inability to tolerate lavage correctly with a preliminary nasal lavage at screening.
* participation in a study with a new molecular entity during the previous four months or any other trial during the previous three months.

Subjects who/with:

* regularly, or on average, drink more than four units of alcohol per day.
* are in receipt of prescribed or over the counter medication (including herbal remedies and dietary supplements) within 14 days of the first dose of test article and for the duration of the trial (with the exception of paracetamol up to 2g daily). In particular, all antihistamines, chromoglycate and steroids are prohibited during this period.
* inability to communicate well with the investigator (i.e., language problem, poor mental development or impaired cerebral function).
* have donated 450 mL or more blood within the previous 12 weeks.
* clinical features suspicious of tuberculosis - weight loss, haemoptysis pyrexia, purulent sputum, previous abnormal chest X-ray will be excluded from the study.
* clinical evidence of autoimmune disease.
* with allergy to seafood or any of the excipients in the study drug formulation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in levels of cytokines in nasal lavage fluid compared with dosing with placebo. | Period 1, day 0. Period 2, day 14
  Change in levels of cytokines (TNF-alfa, IFN-gamma, IL-1b, IL-4 IL5, IL, 6, IL-8, IL-10 and IL-13) in nasal lavage fluid compared to dosing with placebo.

SECONDARY OUTCOMES:
Changes in levels of cytokines in nasal lavage fluid compared with dosing with active control. | Day0, day 14,day 28.
  Changes in levels (maximum concentration) of TNF-alfa, IFN-gamma, IL-1b, IL-4, IL5, IL-6, IL-8, IL-10 and IL-13 in nasal lavage samples following intranasal dosing with cmp compared to lipopolysaccharide active control.
Change from baseline. | Day 0, day 14, day 28
  The total eosinophil counts and cysteinyl leukotriene concentration in nasal lavage fluid following intranasal dosing with cmp.
  Total nasal symptom scores at 4 and 8-hours following intranasal dosing with cmp.
Safety check. | Day0, day14, day 28.
  Safety will be assessed using the adverse events, vital signs and nasal acoustic rhinometry following dosing with cmp versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Professor, Principal Investigator — Aarhus University, School of Public Health, Dept of Environmental & Occupational Medicine
Locations (1):
- Aarhus University, School of Public Health, Dept. of Environmental & Occupational Medicine, Aarhus C, Denmark